CLINICAL TRIAL: NCT05346458
Title: A Single Centre, Prospective, Feasibility Study of the iKOs™ Coronary Pressure and Flow Rapid-exchange Microcatheter and iKOr™ Console in Patients With Coronary Heart Disease Undergoing Coronary Physiology Investigations
Brief Title: Measuring Blood Flow in Heart Vessels With a New Fibre Optic Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Echopoint Medical Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 305877
Record Dates: First submitted 2022-03-09; First posted 2022-04-26 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Coronary Stenosis; Coronary Microvascular Disease
Keywords: Heart; Microcatheter; Fibreoptic
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Microvascular Angina

STUDY DESIGN:
Intervention Model Description: A single centre, prospective, feasibility study of the iKOs™ coronary pressure and flow rapid-exchange microcatheter and iKOr™ console in patients with coronary heart disease undergoing coronary physiology investigations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra coronary rapid-exchange iKOs microcatheter intervention (Experimental): Patients with coronary heart disease and undergoing coronary physiology investigations (pressure wire measurements) will have additional coronary pressure and flow measurements using the iKOs rapid-exchange microcatheter and iKOr console.
  Interventions: Device: Intra coronary rapid-exchange iKOs microcatheter intervention

INTERVENTIONS:
Device: Intra coronary rapid-exchange iKOs microcatheter intervention — Patients planned for an invasive coronary physiology (pressure-wire) study and who meet the inclusion criteria and none of the exclusion criteria can be enrolled. Participants will undergo preparation for their clinical procedure (angiogram with pressure wire study) in the normal manner. Arterial cannulation will be performed via the radial or femoral artery) under local anaesthesia. The sheath will be inserted and a pre-procedure blood sample taken for Troponin T level. A coronary angiogram will be performed as per standard clinical practice prior to cannulating the coronary artery to be studied. The pressure studies will be performed sequentially, first with a pressure wire before using the iKOs™ microcatheter. Following withdrawal of the iKOs™ microcatheter. A pressure wire assessment is repeated after the microcatheter is withdrawn. The case will then proceed as clinically indicated. Post-procedure the participant will be managed according to standard clinical practice.
  Other Names: iKOs Microcatheter

SUMMARY:
The purpose of this investigation is to see if the newly developed "iKOs™ microcatheter" can safely and accurately measure flow and pressure within the heart arteries of 10 patients undergoing angiogram and pressure wire tests.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks and benefits, participants who provide written consent will be screened to make sure they fulfil the study entry requirements. Those who are assessed as eligible will undergo baseline assessments and preparation for their angiogram.

Once enrolled they will undergo coronary angiography at the start of their clinical procedure. The angiogram will be examined by the Investigator and a decision made if the target vessel is suitable for a pressure wire study and insertion of the investigational device. If the investigator confirms that the participant remains eligible and the study part can go ahead, the participant will proceed to undergo the investigation with the iKOs microcatheter.

The study assessments will be performed through the right radial artery (preference) under local anaesthesia. A sheath will be inserted and a pre-procedure blood sample taken for Troponin T level. A pressure study will then be performed, initially with a pressure wire before using the iKOs™ microcatheter. Both will be performed before and after hyperaemia. Following withdrawal of the iKOs™ microcatheter, a pressure wire assessment is then repeated after the microcatheter is withdrawn. The case will then proceed as clinically indicated. The whole procedure should take about 30-45 minutes. Post-procedure the participant will be managed according to standard clinical practice.

The participant will be discharged home, usually about 4 hours after the end of the procedure. A troponin blood test and ECG will be repeated before they are discharged.

Follow up telephone calls to assess for any complications of the procedure will be made within the first 7 days and again between 6 and 8 weeks after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent
* >18 years old
* Have a clinical diagnosis of coronary artery disease
* Undergoing further assessment of a coronary artery with a pressure wire study

Exclusion Criteria:

General

* Previous coronary artery bypass grafting.
* Non/ST-elevation myocardial infarction as indication for angiography.
* Ongoing evidence of ischaemia at rest.
* Severe renal impairment (GFR <25).
* Severe anaemia (Hb <10).
* Heparin allergy.
* Atrial fibrillation.
* Contraindication to adenosine.
* Pregnant or lactating; or female of childbearing potential.
* Participation in other interventional studies.

Additional exclusion criteria at Angiogram:

* Critical coronary artery stenosis in the vessel which is to be studied (>90%).
* Left main stem coronary disease causing a >50% stenosis.
* Triple vessel coronary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of the iKOr system in measuring temperature change (flow) in patients with coronary artery disease undergoing physiology investigations | Measured immediately prior to adenosine administration (baseline), and during adenosine administration (hyperaemia).
  A change in thermal transit time measured by the iKOr system

SECONDARY OUTCOMES:
To assess the safety of the iKOs microcatheter in patients undergoing angiography and pressure wire assessment | Measured at procedure, at 4 hrs post procedure, at 1 week post procedure and 8 weeks post procedure
  The number of major adverse cardiac events or patient deaths
To assess the safety of the iKOs microcatheter procedure | Measured at procedure, 4 hrs post procedure, at 1 week post procedure and 8 weeks post procedure
  The number of procedural complications related to the device (operator observed vessel spasm, vascular complications, bleeding)
To assess the effect of the iKOs microcatheter on cardiac injury | Troponin T measurement at procedure start and 4 hrs post procedure
  The change in Troponin levels
To assess the effect of the iKOs microcatheter on TIMI (Thrombolysis In Myocardial Infarction) flow | TIMI flow measured immediately prior to insertion of iKOs microcatheter and on removal of the iKOs microcatheter
  The change in TIMI (Thrombolysis In Myocardial Infarction) flow

OTHER OUTCOMES:
To examine the quality of the temperature recordings | Measured from just prior to adenosine administration (baseline), and during adenosine administration (hyperaemia).
  The number of complete temperature measurement recordings and the number of interpretable temperature waveforms
To examine ease of use of the iKOs microcatheter | Measured at procedure - the time taken from insertion of iKOs microcatheter into guide cath to removal of iKOs microcatheter from guide cath
  Time taken for deployment of the microcatheter

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mathur, Principal Investigator — Queen Mary University of London
Locations (1):
- St Bartholomew's Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No